CLINICAL TRIAL: NCT04654494
Title: Colorectal Cancer in Crohn's Disease: Long Term Outcomes of Different Surgical Procedures
Brief Title: Colorectal Cancer in Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giuseppe Sigismondo Sica, Associate Professor, Head of Department, University of Rome Tor Vergata
Other Study IDs: REGISTROSPERIMENTAZIONI120/20
Record Dates: First submitted 2020-11-29; First posted 2020-12-04 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Crohn Disease; Colorectal Cancer; Inflammatory Bowel Diseases
Keywords: colorectal surgery
MeSH Terms: conditions — Crohn Disease; Colorectal Neoplasms; Inflammatory Bowel Diseases | interventions — Proctocolectomy, Restorative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chron's disease patients with colorectal cancer: This group of patients with Chron's disease have been diagnosed with colorectal cancer and treated surgically
  Interventions: Procedure: Total proctocolectomy; Procedure: Total colectomy; Procedure: Segmental colectomy

INTERVENTIONS:
Procedure: Total proctocolectomy — excision of the whole large bowel including colon and rectum and end ileostomy fashioning
Procedure: Total colectomy — excision of the colon with preservation of the rectum
Procedure: Segmental colectomy — excision of a segment of colon

SUMMARY:
Retrospective multicentre study. All patients with a diagnosis of Crohn's disease (CD) and operated for colorectal cancer (CRC) between 01/01/2010 and 01/01/2020 will be included in the dataset.

Data will include preoperative, intraoperative and postoperative variables, with long term follow up when feasible.

The study will focus on a comparison between patients treated with total proctocolectomy (TPC) and patients treated with subtotal colectomy (STC) or segmental resection (SR).

Primary endpoints will be oncologic outcomes, postoperative morbidity and mortality. Secondary endpoints include quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of Crohn's disease and concomitant primary colorectal cancer who underwent surgery in an expert centre between 01/01/2010 and 01/01/2020

Exclusion Criteria:

* Patients who underwent non-oncologic segmental resection will be excluded from outcome analysis.
* Patients with known genetic colorectal cancer syndromes (eg. Familial Adenomatous Polyposis, Hereditary Non-Polyposis ColoRectal Cancer Syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn's disease complicated by occurrence of colorectal cancer, treated surgically between 01/2010 and 01/2020
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years
  percentage of patients alive
disease free survival | 5 years
  percentage of patients disease free

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Tor Vergata, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No